CLINICAL TRIAL: NCT06364176
Title: Targeting Inflammation With Losartan to Improve Response to Modulator Therapy in Cystic Fibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00149479
Record Dates: First submitted 2024-03-06; First posted 2024-04-15 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis
Keywords: losartan
MeSH Terms: conditions — Cystic Fibrosis | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Losartan (Experimental): Losartan 25mg twice daily for one week followed by 50mg twice daily through week 12.
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): Placebo twice daily through week 12
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — Treatment with losartan through week 12
  Arms: Losartan
Drug: Placebo — Treatment with placebo through week 12
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test use of losartan in those with cystic fibrosis (CF) on modulator therapy. The main question it aims to answer is if treatment with losartan improves response of the CF transmembrane conductance regulator (CFTR) channel to modulator therapy.

Participants will be asked take losartan or placebo for twelve weeks and will have changes in sweat chloride levels measured as a marker of CFTR function.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, parallel group clinical trial in those those with CF on elexacaftor/tezacaftor/ivacaftor to determine if treatment with losartan improves response to modulator therapy using sweat chloride as an marker of CFTR function.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of cystic fibrosis
* Age 12 years and older
* Stable use of elexacaftor/tezacaftor/ivacaftor for 90 days prior to enrollment
* Sweat chloride concentration 50 mmol/L or greater while on elexacaftor/tezacaftor/ivacaftor

Exclusion Criteria:

* Prior lung transplant
* BMI <18
* CF pulmonary exacerbation requiring hospitalization or intravenous antibiotics in the preceding 30 days
* Systemic corticosteroid or regular non-steroidal anti-inflammatory use in the preceding 30 days
* Chronic use of angiotensin receptor blockers or angiotensin converting enzyme inhibitors
* Concomitant use of medications known to interact with losartan, including aliskiren
* Chronic renal insufficiency (creatinine clearance <45 ml/min)
* Pregnancy or lactation
* Inability or unwillingness to comply with approved contraceptive method during the study period (females of childbearing age)
* In the opinion of the investigator any severe or acute or chronic condition or laboratory abnormality that may increase the risk associated with trial participation or make the participant inappropriate for enrollment
* Participation in another interventional trial that, in the opinion of the investigator, has the potential to affect the primary outcome

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Sweat chloride | Baseline through week 12
  Change in sweat chloride concentration

SECONDARY OUTCOMES:
Lung function - absolute | Baseline through week 12
  Absolute change in percent predicted forced expiratory volume in one second (ppFEV1)
Lung function - relative | Baseline through week 12
  Relative change in ppFEV1
Transforming growth factor (TGF)-beta1 - airway | Baseline through week 12
  Change in nasal fluid levels of TGF-beta1
TGF-beta1 - systemic | Baseline through week 12
  Change in plasma levels of TGF-beta1
Inflammatory mediators - airway | Baseline through week 12
  Change in concentration nasal fluid levels of inflammatory mediators (interleukin-1beta, interleukin-8, tumor necrosis factor-alpha)
Inflammatory mediators - systemic | Baseline through week 12
  Change in plasma levels of inflammatory mediators (interleukin-1beta, interleukin-8, tumor necrosis factor-alpha)
CFQ-R | Baseline through week 12
  Change in CF questionnaire revised (CFQ-R); scale 0-100 with higher scores indicating better quality of life
Adverse events | Baseline through week 12
  Cumulative incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bengtson, MD, MSc, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes